CLINICAL TRIAL: NCT07377916
Title: A Prospective, Single-Arm, Exploratory Clinical Study of SHR-A1811 Combined With Pertuzumab as Second-Line Therapy in Patients With HER2-Altered Advanced Non-Small Cell Lung Cancer
Brief Title: Clinical Study of SHR-A1811 Combined With Pertuzumab as Second-Line Therapy in Patients With HER2-Altered Advanced NSCLC
Acronym: NSCLC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Maoming People's Hospital (Other); Peking University Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Jianxing He, Guangzhou Medical University Affiliated First Hospital National Respiratory Research Center, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-2025-235-02
Record Dates: First submitted 2025-12-02; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1811 combined with pertuzumab (Experimental): Intravenous infusion，Q3 week, SHR-A1811 combined with pertuzumab
  Interventions: Drug: SHR-A1811

INTERVENTIONS:
Drug: SHR-A1811 — Intravenous infusion, q3 week, SHR-A1811 combined with pertuzumab

SUMMARY:
The study enrolled patients with advanced or metastatic NSCLC harboring HER2 mutations, amplification, or overexpression who had progressed after ≥1 prior lines of anticancer therapy. After enrollment, participants received treatment with rezetamab plus pertuzumab until disease progression, intolerable toxicity, withdrawal of consent, or other conditions requiring treatment discontinuation.

DETAILED DESCRIPTION:
Patients who meet the following criteria are enrolled:

Aged 18-75 years Histologically or cytologically confirmed advanced or metastatic non-small cell lung cancer (NSCLC) (AJCC 9th edition) Pathologically documented HER2 mutation, amplification, or overexpression Received ≥1 prior line of systemic anti-cancer therapy for advanced/metastatic disease Received SHR-A1811 combined with pertuzumab

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years
* Histologically or cytologically confirmed advanced or metastatic non-small cell lung cancer (NSCLC) (AJCC 9th edition)
* Pathologically documented HER2 mutation, amplification, or overexpression
* Received ≥1 prior line of systemic anti-cancer therapy for advanced/metastatic disease
* There is at least one measurable lesion according to RECIST V1.1 criteria
* ECOG score of 0 or 1.
* The expected survival is ≥12 weeks

Exclusion Criteria:

* There are untreated or active central nervous system (CNS) tumor metastases
* Has unresolved toxicities from previous anticancer therapy, defined as toxicities not yet resolved to NCI-CTCAE version 5.0 grade ≤ 1.
* Pleural, ascites, or pericardial effusion requiring intervention occurred within 14 days prior to initial administration
* Systemic antitumor therapy was performed 4 weeks prior to study initiation
* Subjects who have previously received HER2-targeted therapy (excluding pan-HER tyrosine kinase inhibitors) or antibody-drug conjugates with a topoisomerase I inhibitor payload.
* Use of strong CYP3A4, CYP2D6, P-gp, or BCRP inhibitors or inducers within less than 5 drug half-lives prior to the first dose.
* Has active infection requiring systemic treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) by investigator assessment | Until progression, assessed up to approximately 2 years

SECONDARY OUTCOMES:
Objective Response Rate （ORR） | Two years after the last subject was enrolled in the group
Overall Survival (OS) | Until death, assessed up to approximately 3 years
Disease Control Rate (DCR) | Two years after the last subject was enrolled in the group
Duration of Response (DOR) | Two years after the last subject was enrolled in the group
AE | until to 90 days after the last dose，assessed up to approximately 3 years

IPD SHARING:
Plan to Share IPD: No